CLINICAL TRIAL: NCT00573131
Title: A Randomized Study of the Efficacy and Safety of OncoGel™ Treatment as an Adjunctive Therapy to Systemic Chemotherapy and Concurrent External Beam Radiation Prior to Surgery in Subjects With Localized or Loco-regional Esophageal Cancer
Brief Title: Efficacy and Safety of OncoGel™ Added to Chemotherapy and Radiation Before Surgery in Subjects With Esophageal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: OncoGel did not show any impact on overall tumor response
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR016-CLN-pro003
Record Dates: First submitted 2007-12-11; First posted 2007-12-13 (Estimated); Results first posted 2014-05-16 (Estimated); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Esophageal Cancer; Adenocarcinoma of the Esophagus; Squamous Cell Carcinoma
Keywords: Esophageal cancer; Localized esophageal cancer; Operable esophageal cancer; Loco-regional esophageal cancer; Esophagectomy; Phase 2; Paclitaxel; Tumor; Local; Chemotherapy; radiation therapy; surgery; OncoGel; Squamous cell carcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus; Carcinoma, Squamous Cell; Neoplasms; Esophageal Squamous Cell Carcinoma | interventions — Cisplatin; Fluorouracil; Radiotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): OncoGel, radiation therapy and systemic chemotherapy (cisplatin plus 5-FU) prior to surgical resection.
  Interventions: Drug: OncoGel (Paclitaxel gel); Drug: cisplatin; Drug: 5-FU; Radiation: radiation therapy; Procedure: esophageal resection
- Group 2 (Active Comparator): Radiation therapy and systemic chemotherapy (cisplatin plus 5-FU) prior to surgical resection.
  Interventions: Drug: cisplatin; Drug: 5-FU; Radiation: radiation therapy; Procedure: esophageal resection

INTERVENTIONS:
Drug: OncoGel (Paclitaxel gel) — 6.3 mg/mL tumor volume, injected into the esophagus during endoscopy, once, before starting chemoradiotherapy
  Arms: Group 1
Drug: cisplatin — 75 mg/m2 IV (in the vein) once on Day 1 and Day 29
Drug: 5-FU — 1000 mg/m2/day, IV (in the vein) for 4 days (96 hours) for two cycles starting on Day 1 and Day 29
Radiation: radiation therapy — 50.4 Gy, given in 28 treatments, once per day for 5 1/2 weeks
Procedure: esophageal resection — Removal of esophagus after completion of chemotherapy and radiation therapy

SUMMARY:
OncoGel is a new experimental drug delivery system that allows the slow continuous release of paclitaxel (an approved intravenous anticancer drug), from a gel (ReGel) over a long period of time. The gel will disappear in 4 to 6 weeks as it releases the paclitaxel.

The protocol is directed towards evaluating the efficacy and safety of paclitaxel delivered as a local, intralesional treatment when used in combination with chemotherapy (cisplatin and 5-FU) and radiation therapy before surgery.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the efficacy of OncoGel given in combination with standard chemotherapy (cisplatin and 5-FU) and radiation therapy in patients with previously untreated, resectable, local or local-regional adenosarcoma or squamous cell carcinoma.

All patients will receive IV cisplatin on Day 1 and Day 29 and IV 5-FU given continuously for 96 hours starting on Day 1 and Day 29. All patients will also receive out-patient radiation therapy for 28 treatments once per day for 5 1/2 weeks starting on Day 1.

Patients randomized to the OncoGel treatment group will have the OncoGel dose injected into their esophageal tumors during an endoscopic procedure just before starting systemic chemotherapy and radiation therapy.

All patients will have CT scans for tumor measurements before starting chemotherapy and 12 weeks later after completion of the radiation therapy and both cycles of chemotherapy.

During the chemotherapy and radiation therapy, physical exams, vital signs, routine blood tests will be performed. Patients will also be asked about their quality of life and ability to swallow.

In-patient surgery will be scheduled 4 to 6 weeks after completion of chemotherapy and radiation therapy. The resected esophagus and lymph nodes will be evaluated for the presence of residual tumor.

Patients will be followed at months 4, 5, 6, and then every 3 Months thereafter for survival and esophageal cancer status and treatment until the last patient enrolled has completed their Month 12 visit.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed squamous cell carcinoma or adenocarcinoma of the esophagus. Stage T2-T3, N any, M0 (no evidence of disseminated cancer except regional involvement which may be designated as "M1a"). No evidence of metastatic disease
2. Medically able to tolerate major abdominal and/or thoracic surgery
3. Able to undergo EUS procedure and pass EUS probe through esophageal lumen
4. Able to receive concurrent systemic chemotherapy (cisplatin and 5-FU) and RT
5. Clinical management plan includes esophagectomy after completion of two courses of chemoradiation therapy
6. Karnofsky Performance Status of ≥ 60
7. Minimum life expectancy of 4 months
8. Hematologic function

   * Absolute neutrophil count (ANC) ≥ 1500/mm3
   * Platelet count ≥ 100,000/mm3
   * Hemoglobin ≥ 9 g/dL
9. Hepatic function:

   * Total bilirubin < 1.5 X upper limit of normal (ULN)
   * AST and ALT < 3 X ULN
   * Albumin ≥ 3.0 g/dL or ≥ 2.0 g/dL if the lower level is considered by the investigator to be due to nutritional depletion
10. Serum creatinine < 1.5 mg/dL and/or creatinine clearance ≥ 65 mL/min
11. ≥ 18 years old
12. If female, must be non-pregnant, nonlactating, of non-childbearing potential, or using adequate birth control
13. Capable of understanding and agreeing to fulfill the requirements of the protocol
14. Sign the IRB/EC approved consent form

Exclusion Criteria:

1. History of anaphylaxis to planned CT contrast agent
2. Prior esophageal stent insertion, laser, or photodynamic therapy
3. Prior chest RT or major esophageal surgery
4. Any prior receipt of cytotoxic chemotherapeutic agents
5. Prior receipt of other cancer treatments (ie, Chelation therapy), vaccines, or biological response modifiers/growth factors (ie, GM-CSF, IL-2) within the past 4 weeks.
6. Prior malignancy unless disease free for ≥ 3 years. Note: basal cell/squamous carcinoma of the skin, in situ cervical or breast carcinoma, or superficial transitional cell bladder carcinoma will be allowed. Subjects with a history of low risk prostatic carcinoma (ie, clinical stage 1 or 2a, Gleason score < or = 6 and PSA <10 ng/mL at diagnosis) will be allowed
7. Significant currently active systemic diseases including uncontrolled diabetes, severe heart disease (New York Heart Association Class III or IV), uncontrolled hypertension, myocardial infarction within 3 months, severe bronchial obstruction, uncontrolled seizure disorder, or peripheral neuropathy greater than CTCAE grade 1
8. Allergies to any of the active or inactive components of OncoGel (ie, allergies to degradable PLGA [poly(lactide-co-glycolide) sutures])
9. Receipt of an investigational drug or device within 30 days prior to signing informed consent
10. Any medical condition or other circumstance that, in the Investigator's opinion, would prevent completion of the study, interfere with analysis of the study results, or potentially adversely affect subject safety
11. Known esophageal varices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2008-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirk D Fowers, PhD, Study Director — Boston Scientific Corporation
Locations (20):
- United States (8):
  - University of California San Diego, San Diego, California
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Baylor University Medical Center, Dallas, Texas
  - Digestive Health Specialists of Tyler, Texas, Tyler, Texas
- Czechia (5):
  - University Hospital Brno, Brno
  - Hospital Jablonec nad Nisou, Jablonec nad Nisou
  - University Hospital Olomouc, Olomouc
  - University Hospital Motol, Prague
  - Massaryk's Hospital in Usti nad Labem, Ústí nad Labem
- India (5):
  - Kidwai Memorial Institute of Oncology, Bangalore, Karnataka
  - Amrita Institute of Medical Sciences, Kochi, Kerala
  - Bombay Hospital & Medical Research Centre, Mumbai, Maharashtra
  - Deenanath Mangeshkar Hospital, Erandwane, Pune
  - Meenakshi Mission Hospital and Research Centre, Madurai, Tamil Nadu
- Poland (2):
  - Samodzielny Publiczny Szpital Kliniczny, Lublin
  - Samodzielnego Publicznego Szpitala Klinicznego, Szczecin

REFERENCES:
- [Derived] DeWitt JM, Murthy SK, Ardhanari R, DuVall GA, Wallner G, Litka P, Daugherty C, Fowers K. EUS-guided paclitaxel injection as an adjunctive therapy to systemic chemotherapy and concurrent external beam radiation before surgery for localized or locoregional esophageal cancer: a multicenter prospective randomized trial. Gastrointest Endosc. 2017 Jul;86(1):140-149. doi: 10.1016/j.gie.2016.11.017. Epub 2016 Nov 24. PMID 27890801

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from 21 Jan 2008 through 05 Nov 2010 at 20 centers in 5 countries (United States, India, Poland, Czech Republic and Belgium).
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 72 | 65
Completed | 62 | 57
Not Completed | 10 | 8
Not completed — Withdrawal by Subject | 10 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 72 | 65 | 137
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 55 | 48 | 103
  >=65 years | 17 | 17 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (7.2) | 57.6 (10.9) | 58.0 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 40
  Male | 53 | 44 | 97
Region of Enrollment [Number; unit: participants]
  United States | 13 | 9 | 22
  Czech Republic | 14 | 11 | 25
  Poland | 8 | 9 | 17
  Belgium | 0 | 1 | 1
  India | 37 | 35 | 72

OUTCOME MEASURES:

1. Primary Outcome: Overall Tumor Response at the Primary Tumor Site Based on Measurement of Primary Tumor Volume (Excluding Involved Lymph Nodes) by Spiral CT
Description: Per the Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and by Spiral CT assessment:
  Complete Response (CR) is the disappearance of all target lesions; Partial Response (PR) is a >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Screening and Week 12
Population: Subjects who received at least one treatment with OncoGel, systemic chemotherapy or external beam radiation therapy were included for analysis of efficacy.
Measure: Number; unit: percentage of patients
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 72 | 65
percentage of patients | 12.5 | 20.0

ADVERSE EVENTS:
Time Frame: Adverse events were collected through the 12 week Assessment Period
Description: Serious adverse events were collected through the first 30 days after the Week 12 visit
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 30/72 | 20/65
Other Adverse Events (participants affected / at risk) | 67/72 | 55/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=72) | Group 2 (N=65)
Leukopenia (Blood and lymphatic system disorders) | 3 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Granulocytopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 4
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Aphagia (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 4
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Oesophageal perforation (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 3 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Chest pain (General disorders) | 1 | 0
Disease progression (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lung abscess (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Facial palsy (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Hemiplegia (Nervous system disorders) | 0 | 1
Syncope vasovagal (Nervous system disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Arterial thrombosis limb (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=72) | Group 2 (N=65)
Anaemia (Blood and lymphatic system disorders) | 6 | 7
Leukopenia (Blood and lymphatic system disorders) | 17 | 8
Neutropenia (Blood and lymphatic system disorders) | 6 | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 12 | 8
Abdominal pain (Gastrointestinal disorders) | 8 | 5
Constipation (Gastrointestinal disorders) | 14 | 9
Diarrhoea (Gastrointestinal disorders) | 11 | 10
Dysphagia (Gastrointestinal disorders) | 7 | 9
Nausea (Gastrointestinal disorders) | 24 | 11
Odynophagia (Gastrointestinal disorders) | 6 | 4
Oesophagitis (Gastrointestinal disorders) | 5 | 3
Vomiting (Gastrointestinal disorders) | 13 | 15
Asthenia (General disorders) | 3 | 4
Chest pain (General disorders) | 11 | 6
Fatigue (General disorders) | 11 | 9
Mucosal inflammation (General disorders) | 5 | 5
Pyrexia (General disorders) | 13 | 12
Weight decreased (Investigations) | 14 | 12
Anorexia (Metabolism and nutrition disorders) | 7 | 9
Dehydration (Metabolism and nutrition disorders) | 5 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 7
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Dizziness (Nervous system disorders) | 4 | 4
Insomnia (Psychiatric disorders) | 6 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 13
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Hypotension (Vascular disorders) | 1 | 5

LIMITATIONS AND CAVEATS:
Study prematurely terminated due to lack of efficacy in primary endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days